CLINICAL TRIAL: NCT07389434
Title: Feasibility, Safety, Cost-effectiveness, and Environmental Impact of Reprocessed Ablation Catheters in Pulmonary Vein Isolation
Brief Title: Feasibility, Safety, Cost-effectiveness, and Environmental Impact of Reprocessed Ablation Catheters in PVI
Acronym: RE-USE PVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Ivan Zeljkovic, Principal Investigator and Head of Diagnostic and Therapeutic Department for Cardiac Electrostimulation and Electrophysiology, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/1024-3
Record Dates: First submitted 2026-01-09; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Catheter Ablation; Electroporation; Catheter Reprocessing; Cost-Benefit Analysis; Medical Waste; Environmental Impact
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective, randomized, controlled non-inferiority trial with a parallel-group design, comparing resterilized (reprocessed) and new electroporation ablation catheters used for pulmonary vein isolation in patients with atrial fibrillation. Participants will be randomly assigned to two groups, with one group undergoing ablation using new catheters and the other using resterilized catheters, while the procedural protocol will be identical in both groups. The primary endpoint is procedure duration, expressed in minutes. Secondary endpoints include catheter functionality, fluoroscopy time and radiation dose, peri- and post-procedural complications, procedural safety, procedural costs, and assessment of environmental impact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reprocessed Catheter (Experimental) (Experimental): Participants will undergo pulmonary vein isolation using a reprocessed electroporation ablation catheter. The catheter has undergone validated cleaning, re-sterilization, and functional testing in accordance with applicable regulatory and safety standards. Procedural technique, energy delivery protocol, and peri-procedural management will be identical to those used in the comparator arm.
  Interventions: Procedure: Participants will undergo pulmonary vein isolation using pulsed field ablation (PFA). The intervention consists of the use of either a reprocessed electroporation ablation catheter or a new electropor
- New Catheter (Active Comparator) (Active Comparator): Participants will undergo pulmonary vein isolation using a new electroporation ablation catheter. Procedural technique, energy delivery protocol, and peri-procedural management will be identical to those used in the experimental arm.
  Interventions: Procedure: Participants will undergo pulmonary vein isolation using pulsed field ablation (PFA). The intervention consists of the use of either a reprocessed electroporation ablation catheter or a new electropor

INTERVENTIONS:
Procedure: Participants will undergo pulmonary vein isolation using pulsed field ablation (PFA). The intervention consists of the use of either a reprocessed electroporation ablation catheter or a new electropor — This intervention involves pulmonary vein isolation performed with ablation catheter that is either new or reprocessed. The reprocessed catheter has undergone validated cleaning, resterilization, and functional testing in accordance with regulatory and safety standards prior to reuse. The key distinguishing feature of this intervention is the comparison of reprocessed versus new single-use catheters, while all other procedural aspects, including operator technique, energy delivery protocol, and peri-procedural care, are standardized and identical between groups.

SUMMARY:
This study evaluates whether re-sterilized (reprocessed) ablation catheters are as effective and safe as new ablation catheters when used for pulmonary vein isolation in patients with atrial fibrillation. Adult patients scheduled for catheter ablation will be randomly assigned to undergo the procedure using either a new catheter or a re-sterilized catheter, with identical procedural techniques applied in both groups. The study will compare procedural efficiency, safety, costs, and environmental impact between the two approaches. The results may support more sustainable and cost-effective use of medical devices in cardiac electrophysiology.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled non-inferiority trial comparing re-sterilized (reprocessed) and new ablation catheters for pulmonary vein isolation in patients with atrial fibrillation. The study will be conducted at University Hospital Dubrava, a high-volume tertiary center for cardiac electrophysiology.

Patients scheduled for pulmonary vein isolation will be randomized in a 1:1 ratio using a computer-generated sequence to undergo ablation with either a new or a re-sterilized catheter. All procedures will be performed by experienced electrophysiologists in accordance with standard institutional practice.

Procedure duration will be measured from transseptal puncture to completion of ablation of all pulmonary veins. Additional procedural parameters related to ablation delivery, including duration and number of energy applications, total ablation time, and other procedural timing characteristics, will also be recorded. Fluoroscopy time and radiation dose, expressed as dose-area product (DAP), will be recorded automatically.

Catheter performance will be assessed based on achievement of complete pulmonary vein isolation, the number of energy applications per pulmonary vein, and procedural assessment of catheter integrity, flexibility, and electrical properties.

Procedural safety will be evaluated by monitoring peri-procedural and post-procedural adverse events, including pericardial effusion, stroke, vascular complications, and death. Laboratory markers of inflammation, infection, and hemolysis will be obtained at predefined time points before and after the procedure. Blood cultures will be collected after the procedure to assess potential infectious complications.

Patients will be followed clinically during hospitalization and after discharge through telephone contact and routine outpatient visits.

Economic evaluation will include direct procedural costs, catheter costs, and re-sterilization costs. Environmental impact will be assessed based on medical waste generation and estimated carbon footprint associated with catheter use.

Re-sterilization of ablation catheters will be performed according to the validated internal protocol of University Hospital Dubrava, which has been used in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Paroxysmal or persistent atrial fibrillation documented by ECG or Holter ECG monitoring
* Indication for pulmonary vein isolation according to current clinical guidelines
* Written informed consent

Exclusion Criteria:

* Severe valvular heart disease
* Significant structural heart disease that precludes pulsed field ablation (PFA)
* Pregnancy or breastfeeding
* Life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vein Isolation Procedure Duration | From the start of the index ablation procedure until its completion.
  Procedure duration, expressed in minutes, measured from transseptal puncture to completion of ablation of all pulmonary veins. Additional procedural parameters, including duration of individual procedural segments, total ablation time, number and duration of energy applications, and other time-related procedural characteristics, will also be recorded.

SECONDARY OUTCOMES:
Procedural Catheter Performance Parameters | From the start of the index ablation procedure until its completion
  Catheter functional performance assessed by successful pulmonary vein isolation, number of energy applications per pulmonary vein, total ablation time, and procedural assessment of catheter integrity and flexibility.
Medical Waste Generated Per Procedure | Periprocedural
  Amount of medical waste generated per ablation procedure, expressed in kilograms.
Fluoroscopy Time | From the start of the index ablation procedure until its completion
  Total fluoroscopy time, expressed in minutes, recorded during the ablation procedure.
Radiation Dose (Dose-Area Product) | From the start of the index ablation procedure until its completion
  Radiation exposure expressed as dose-area product (DAP), automatically recorded during the ablation procedure.
Incidence of Peri- and Post-Procedural Complications | Up to 30 days following the index ablation procedure
  Number of participants with peri-procedural and post-procedural complications, including pericardial effusion, stroke, vascular complications, and death.
Direct Procedural Costs Per Patient | Periprocedural
  Direct procedural costs per patient, including catheter cost, procedure-related costs, and re-sterilization costs, expressed in local currency.
Estimated Carbon Footprint Per Procedure | From the start of the index ablation procedure until its completion.
  Estimated carbon footprint associated with the ablation procedure and catheter use, expressed in CO₂-equivalent units.

CONTACTS AND LOCATIONS:
Locations (1):
- UH Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as no formal data-sharing plan has been established for this study.